CLINICAL TRIAL: NCT01400464
Title: Study the Link Between Steroids Pharmacokinetics and the Response to Prednisone Therapy in Giant Cell Arteritis
Brief Title: Steroids Pharmacokinetics and the Response to Prednisone Therapy in Giant Cell Arteritis
Acronym: PREDICORT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-004896-23
Record Dates: First submitted 2011-07-21; First posted 2011-07-22 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Giant Cell Arteritis
Keywords: Giant Cell Arteritis; prednisone; pharmacokinetics
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Prednisone therapy and pharmacokinetic — Prednisone therapy delivered in accordance with a 10 to 18 month pre-defined schedule. Pharmacokinetic and pharmacogenetic tests at 14 or 28 days. Monthly visit for the first 6 month, then every 8 weeks months thereafter for the remainder of the study with standard biologic monitoring , physical exam and medical and medication history .Also, participants will be asked to complete several questionnaires to assess quality of life and observance to therapy. Participants may have additional study visits if a disease flare or disease-related complications occur during the study.

SUMMARY:
The factors underlying the large interindividual variability in response to glucocorticoids in Giant Cell Arteritis are poorly understood. The investigators hypothesize that a part of this variability is related to pharmacokinetic factors determined by genetic polymorphism: hepatic clearance involving cytochromes P450 of the subfamily 3A (CYP3A) and drug efflux leukocyte conditioned by P-glycoprotein involved in multidrug resistance drugs (ABCB1). The investigators have designed a multicentric prospective pharmacokinetical and pharmacogenetic cohort study to assess the link between prednisolone clearance and the relapse risk in giant cell arteritis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GCA, meeting at least 3 of the following 5 American College of Rheumatology (ACR) criteria for the diagnosis of GCA:

  1. At least 50 years of age at disease onset
  2. New onset or new type of localized pain in the head
  3. Temporal artery abnormality (i.e., temporal artery tenderness to palpation or decreased pulsation unrelated to arteriosclerosis of cervical arteries)
  4. ESR of greater than 40 mm in the first hour by the Westergren method
  5. Temporal artery biopsy showing vasculitis characterized by a predominance of mononuclear cell infiltration or granulomatous inflammation, usually with multinucleated giant cells
* Corticoid treatment since less than 14 days
* Signed informed consent
* Affiliation to the social security system

Exclusion Criteria:

* Dementia
* Predictable non observance
* Neoplasia since less than 5 years

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-07; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
oral clearance of prednisolone | 2 to 4 weeks after begining prednisolone treatment

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - CHU de CAEN, Caen, Etat
  - Hôpital Cochin-APHP, Paris, Etat
  - Centre Hospitalier Universitaire de Toulouse, Toulouse, Etat
  - CH de Valenciennes, Valenciennes, Etat
  - CHU Avicennes, Bobigny
  - CHU Jean Verdier (AP-HP), Bondy
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - CHU de Lille, Lille
  - Centre Hospitalier Universitaire de Limoges, Limoges
  - CHU de Nantes, Nantes
  - Hôpital Pitié-Salpêtrière-APHP, Paris
  - CHU de Rouen, Rouen